CLINICAL TRIAL: NCT07027683
Title: CMR UNCONCEALED Study
Brief Title: Cardiac Magnetic Resonance for Diagnosing and Guiding Treatment in Concealed Myocardial Rupture
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Mattia Alberti, Dr, University of Pisa
Other Study IDs: CMR UNCONCEALED
Record Dates: First submitted 2024-12-07; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Early Infarct-associated Pericarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Post-MI cardiac MRI

SUMMARY:
looking for the incidence of concealed myocardial rupture in patients with post infarct pericarditis

ELIGIBILITY:
Inclusion Criteria:

* STEMI
* Clinical diagnosis of Early infarct-associated pericarditis

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: STEMI patients with a clinical diagnosis of Early infarct-associated pericarditis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Myocardial rupture | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Pisa, Pisa, Italy